CLINICAL TRIAL: NCT04706481
Title: Archival of Human Biological Samples in CU-Med Biobank
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Ronald C.W. Ma, Professor, Chinese University of Hong Kong
Other Study IDs: CREC 2019.152
Record Dates: First submitted 2020-12-28; First posted 2021-01-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Healthy; Cancer; Heart Diseases; Neurological Diseases or Conditions; Kidney Diseases; Diabetes; Other Disease
Keywords: Biobanking
MeSH Terms: conditions — Neoplasms; Heart Diseases; Kidney Diseases; Diabetes Mellitus; Disease | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 99 Years
Biospecimen Retention: Samples With DNA — Bufft coats, plasma, serum, tissues, pleural effusion, urine and stool, etc
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: Healthy subjects who have provided consent for specimen collection
  Interventions: Procedure: Specimen Collection
- Cancer or Other Diseases: Diseased subjects who have provided consent for specimen collection
  Interventions: Procedure: Specimen Collection

INTERVENTIONS:
Procedure: Specimen Collection — Specimens obtained from surgical, phlebotomy or other non-invasive procedure

SUMMARY:
CU-Med Biobank collaborates with different researchers for collecting and distributing human biospecimens and clinical data for assisting scientific research.

DETAILED DESCRIPTION:
CU-Med Biobank will collect and store high-quality specimens from cancer-related or other diseases. All samples are linked to annotated clinical data from approved consented protocols. This system provides researchers with high- quality biological samples and comprehensive clinical, pathological including molecular/genetic information for their research. This standardized CU-Med Biobank is a pivotal bridge to improve the translation of basic research into clinical applications. These findings will contribute to improve prevention, enhance diagnosis, develop new treatment and eventual cure of diseases.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled subjects that have provided signed consent for the specimens and de-identified data to be collected, stored and distributed.

Exclusion Criteria:

* Subjects without signed informed consent for the specimens and de-identified data to be collected, stored and distributed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The diverse group of biorepositories with focus on normal cohorts and cancer-related or other disease cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2050-12-01 (Estimated); Study Completion 2050-12-01 (Estimated)

PRIMARY OUTCOMES:
To distribute human biospecimens for clinical research | 99 years
  By using the biological samples from CU-Med Biobank, translational studies can be done.
To discover the pathological mechanism of different acute and chronic diseases such as cancer, stroke, heart disease, dementia & diabetes | 99 years
  The relationship between different genome/proteome/bacteriome/virome and various diseases can be revealed, thus leading to a better prognostic and diagnostic outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ching Wan MA, MB BChir, Study Chair — Chinese University of Hong Kong
Locations (1):
- CU-Med Biobank, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Webpage of CU-Med Biobank — https://www.med.cuhk.edu.hk/facilities/cu-med-biobank